CLINICAL TRIAL: NCT01083875
Title: A Double-blind, Randomized, Vehicle-controlled Phase II Study to Determine the Effects of Concomitant Treatment With Amlexanox 0.5% Oral Rinse Solution on Oral Mucositis Associated With Radiation Therapy for Cancer of the Head and Neck Region
Brief Title: Study to Determine the Effects Treatment With Amlexanox 0.5% Oral Rinse Solution on Oral Mucositis Associated With Radiation Therapy for Cancer of the Head and Neck Region
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Access Pharmaceuticals, Inc. (Industry)
Collaborators: Advanced Clinical Research Services, LLC (Other)
Responsible Party: David Nowotnik
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-C-9U01
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Oral Mucositis
Keywords: Radiation; mucositis; head and neck carcinoma; oral rinse; amlexanox; MuGard
MeSH Terms: conditions — Stomatitis; Mucositis | interventions — amlexanox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5% amlexanox oral rinse (Experimental): Patients treated with an oral rinse containing the active 0.5% amlexanox
  Interventions: Drug: amlexanox
- Vehicle (Placebo Comparator): Patients treated with an oral rinse containing no active
  Interventions: Drug: Vehicle rinse

INTERVENTIONS:
Drug: amlexanox — 0.5% amlexanox oral rinse; use 5 ml every 2-3 hours during the awake hours of each day (a minimum of 6 times each day). The liquid was be swirled around the mouth then to be swallowed. Repeated daily until completion of radiation therapy: approximately 7-8 weeks.
  Arms: 0.5% amlexanox oral rinse
Drug: Vehicle rinse — use 5 ml of the vehicle rinse every 2-3 hours during the awake hours of each day (a minimum of 6 times each day). The liquid is be swirled around the mouth then swallowed.
  Other Names: MuGard
  Arms: Vehicle

SUMMARY:
The purpose of this study was to determine the effect of 0.5% amlexanox oral rinse compared to a vehicle control on mucositis-related ulceration and erythema (objective score)and on mucositis-related oral pain (subjective score).

A secondary objective was to evaluate the safety of 0.5% amlexanox oral rinse by determining the frequency of treatment-emergent drug-related adverse events or clinical laboratory abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older;
2. Patient has a histologically documented diagnosis of cancer of the head and neck region;
3. Patient is about to receive a course of radiation therapy (with or without concomitant chemotherapy) with a planned dose of at least 60 Gy over 6-7 weeks, and with planned fields to involve at least 50% of the oral mucosa;

This criterion was amended (Amendment 01 dated August 28, 2000) to read as follows:

3. Amended: Patient is at a high risk of developing radiation-induced mucositis. For the purpose of this study, high-risk patients will be defined as:

1. patients about to receive a course of radiation therapy (with or without concomitant chemotherapy) with a planned dose of at least 60 Gy over 6-7 weeks, and
2. with planned fields to involve at least 40% of the oral and oropharyngeal mucosa visible by direct inspection;

   4. Patient has a Karnofsky Performance Scale (KPS) score of 60% or more;

   5. Patient is willing and able to cooperate with the protocol including rinsing of the oral cavity with the investigational or vehicle oral rinse 6 times per day.

   6. The patient or guardian is capable of providing informed consent.

   7. If female, the subject has undergone a urine pregnancy test with negative results, and has agreed to practice effective methods of contraception for the duration of the study.

   Exclusion criteria
   1. Patient has had previous radiation therapy to the oral mucosa;
   2. Patient is about to receive hyperfractionated radiation therapy;
   3. Patient has active oral H. simplex lesions, oral candidiasis, or oral mucositis due to other disease processes;
   4. Patient has uncontrolled infection;
   5. Patient has HIV, Hepatitis B (HBV) (as measured by HBs-Ag) or Hepatitis C (HCV) infection;
   6. Patient has not recovered from oral toxicity attributable to prior treatment;
   7. Patient has abnormal laboratory values that meet the following criteria:

      * Serum creatinine greater than 2 x upper limit of normal
      * Total bilirubin greater than 3 x upper limit of normal;
      * SGOT greater than 3 x upper limit of normal;
      * LDH greater than 3 x upper limit of normal;
   8. Patient has known sensitivities to any of the study preparation ingredients;
   9. Patient has participated in a clinical research study within the last 30 days prior to enrollment;
   10. Patient is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2000-02; Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of mucositis using the Oral Mucositis Assessment Score | 7 weeks

SECONDARY OUTCOMES:
Frequency of treatment-emergent, drug-related Serious Adverse Events | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Busse, M.D., Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (12):
- United States (12):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - University of Arkansas Medical School, Little Rock, Arkansas
  - Florence Wheeler Cancer Center, Bakersfield, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - ICSL Clinical Studies, Melbourne, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - University of Tennessee, Memphis, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Corpus Christi Cancer Center, Corpus Christi, Texas